CLINICAL TRIAL: NCT06691022
Title: Evaluation of the Effects of Passive Smoking and Parental Stress on Challenging Behaviors in Mentally Retarded Children With Urine Cotinine Levels
Acronym: smoking
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mukaddes Demir Acar, Principal Investigator, Tokat Gaziosmanpasa University
Other Study IDs: TOGU2023
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Smoking Behavior; Special Needs Child
Keywords: smoking; Child's Challenging Behaviour; parents; stres
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smoking: not smoking

SUMMARY:
This research was planned to determine the effect of environmental cigarette smoke exposure and parenting stress level on the severity of challenging behaviors in mentally disabled children

DETAILED DESCRIPTION:
This research was planned to determine the effect of environmental cigarette smoke exposure and parenting stress level on the severity of challenging behaviors in mentally disabled children

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-10 with mental disabilities
* Parents' ability to speak and understand Turkish
* Parents' willingness to participate in the study

Exclusion Criteria:

Children who do not match the age group and do not meet the inclusion criteria

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: special needs child
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The Child's Challenging Behaviour Scale 2 (CCBS-2) | 1 years
  face to face
parent stress scaleparent stress scale parent stress scale Parent's Stress Scale | 1 years
  Face to face
cotinin in urine | 1 years
  urine analysis
sociodemographic questionnaire | 1 years
  face to face

CONTACTS AND LOCATIONS:
Locations (1):
- TURKEY, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
to be specific